CLINICAL TRIAL: NCT05936047
Title: Efficacy of Autologous Bone Marrow Clot as Scaffold for Instrumental Posterior Lumbar Fusion
Brief Title: Bone Marrow Clot for Posterior Lumbar Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVOD.clot
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Spinal Fusion
Keywords: Spine; Spinal fusion; Degenerative diseases; Vertebral bone marrow; Clot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The clotted vertebral bone marrow aspirate (vBMA) will be obtained from vertebral bone marrow aspirate.The vBMA clot contain mesenchymal stem cells (MSCs), growth factors, platelet and osteogenic and anti-inflammatory mediators.
  Interventions: Biological: Vertebral bone marrow clot

INTERVENTIONS:
Biological: Vertebral bone marrow clot — vBMA will be harvested from each patient vertebral pedicle with the preparation of the site for pedicle screw insertion during spinal surgery. After the positioning of pedicle screws, the decompression of the cauda and nerve roots will be achieved with a hemilaminectomy and foraminotomy. vBMA clot will be opposed on the hemi-laminae and transvers process on the contralateral side of the hemilaminectomy. On the hemilaminectomy side, foramino-arthrectomy will be performed to insert the interbody fusion cage if necessary. After aspiration, the vBMA will be clotted and used for surgical procedure. vBMA clot will be applied on each side of the vertebra according to the number of segments to be fused.

SUMMARY:
Bone marrow aspirate (BMA) in association to graft substitutes has long been introduced as a promising alternative to iliac crest bone graft in spinal fusion. However, BMA use is limited by the absence of a standardized technique, of a physical texture and by the possibility of dispersion away from the implant site. Recently, the potential use of a new formulation of BMA, named BMA clot, has been preclinically described. A prospective pilot clinical study designed to assessing the safety and efficacy of autologous vertebral BMA (vBMA) clot as multifunctional bio-scaffold in instrumental posterior lumbar fusion will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18 at the time of surgery
* symptomatic degenerative spine disease needing posterior fusion at the lumbar tract

Exclusion Criteria:

* any form of local or systemic infections, inflammatory or autoimmune disease
* coagulation disorders
* tumor diseases
* alcohol or drug abuse
* pregnancy
* chemotherapeutic drugs that might interfere with bone regeneration processes
* revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Brantigan classification | At baseline (day 0)
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at FUs, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).
Brantigan classification | 3 months
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at FUs, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).
Brantigan classification | 12 months
  Improvement of spinal fusion rate and time in patients treated with vBMA clot associated to bone allograft chips in comparison to bone allograft chips alone, also considering age and gender differences. CT-scan and X-ray, perform pre-operatively and at FUs, will be evaluated basing on Brantigan classification (which ranges from A to E, with E score indicating better SF rate).

SECONDARY OUTCOMES:
Visual Analogue Score | At baseline (day 0)
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Visual Analogue Score | 3 months
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Visual Analogue Score | 12 months
  Visual Analogue Score (which ranges from 0 to 100 with higher scores indicating more severe pain)
Oswestry Disability Index | At baseline (day 0)
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Oswestry Disability Index | 3 months
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
Oswestry Disability Index | 12 months
  Oswestry Disability Index (ODI) (which ranges from 0 to 100 with higher scores indicating more severe disability)
EuroQoL-5L (EQ-5L) | At baseline (day 0)
  EuroQoL-5L (EQ-5L) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)
EuroQoL-5L | 3 months
  EuroQoL-5L (EQ-5L) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)
EuroQoL-5L | 12 months
  EuroQoL-5L (EQ-5L) (set of generic and coherent quality-of-life measures based on patient self-reporting outcomes)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salamanna F, Contartese D, Giavaresi G, Sicuro L, Barbanti Brodano G, Gasbarrini A, Fini M. A Rationale for the Use of Clotted Vertebral Bone Marrow to Aid Tissue Regeneration Following Spinal Surgery. Sci Rep. 2020 Mar 5;10(1):4115. doi: 10.1038/s41598-020-60934-2. PMID 32139727
- [Background] Salamanna F, Contartese D, Nicoli Aldini N, Barbanti Brodano G, Griffoni C, Gasbarrini A, Fini M. Bone marrow aspirate clot: A technical complication or a smart approach for musculoskeletal tissue regeneration? J Cell Physiol. 2018 Apr;233(4):2723-2732. doi: 10.1002/jcp.26065. Epub 2017 Jul 24. PMID 28639702
- [Background] Salamanna F, Contartese D, Borsari V, Pagani S, Barbanti Brodano G, Griffoni C, Ricci A, Gasbarrini A, Fini M. Two Hits for Bone Regeneration in Aged Patients: Vertebral Bone Marrow Clot as a Biological Scaffold and Powerful Source of Mesenchymal Stem Cells. Front Bioeng Biotechnol. 2022 Jan 18;9:807679. doi: 10.3389/fbioe.2021.807679. eCollection 2021. PMID 35118056